CLINICAL TRIAL: NCT04058587
Title: Phase I Dose-escalation Trial of Simmitinib for Patients With Advanced Solid Tumors in Therapeutic Failure
Brief Title: A Phase I Trial of Simmitinib in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOMCL-15-290-201901
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simmitinib tablet (Experimental): The core trial period includes 4-weeks Screening stage (28d), 7-days single administration stage, 4-weeks multiple administration stage (28d), 3-days blood collection stage of PK after multiple administration.
  The starting dose was set at 1mg/d on toxicology data. Dosing will continue uninterrupted for 28 days in multiple administration stage.
  The dose-limiting toxicity (DLT) period assessment will be from the first administration of Simmitinib tablet to the end of the first cycle (35 days).
  Interventions: Drug: Simmitinib

INTERVENTIONS:
Drug: Simmitinib — The core trial period includes 4-weeks Screening stage (28d), 7-days single administration stage, 4-weeks multiple administration stage (28d), 3-days blood collection stage of PK after multiple administration.
  The starting dose was set at 1mg/d on toxicology data. Dosing will continue uninterrupted for 28 days in multiple administration stage.
  The dose-limiting toxicity (DLT) period assessment will be from the first administration of Simmitinib tablet to the end of the first cycle (35 days).
  Other Names: SOMCL-15-290

SUMMARY:
This is an open label, multi-center, phase I study of oral Simmitinib in subjects with advanced solid tumors including gastric cancer.

DETAILED DESCRIPTION:
This is an open label, multi-center, phase I study of oral Simmitinib in subjects with advanced solid tumors including gastric cancer [including gastroesophageal cancer], cholangiocarcinoma, lung squamous cell carcinoma, urothelial transitional cell carcinoma, and estrogen-receptor-positive breast cancer patients [ER+], etc. This phase I study will evaluate the safety, tolerability, pharmacokinetics and the preliminary efficacy of the FGFR/KDR/CSF1R multi-target inhibitor Simmitinib.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the patient obtained before any study-specific procedure；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* Patients with histologically/cytologically confirmed diagnosis of advanced solid tumors refractory to standard therapy or for whom no standard therapy exist;
* Adequate washing period from last anti-tumor therapy;
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1;
* The expected survival time for more than 12 weeks;
* Adequate bone marrow, hepatic, renal, pancreas, and coagulation function, Blood phosphorus and calcium in the normal range.

Exclusion Criteria:

* Prior treatment with selective FGFR inhibitors or multi-target kinase Inhibitors with FGFR as the main target;
* Unrecovered from any drug-related adverse event to grade ≤ 1 according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.3.0 derived from any previous anti-tumor treatment, excluding alopecia, Pigmentation, or other toxicity with little safety risk for subjects;
* Active Central Nervous System (CNS) metastases (brain or leptomeningeal metastases, etc.);
* Any other history of malignancy within 3 years;
* Congenital coagulation abnormalities. Active bleeding or previous history of massive bleeding (>30ml within 3 months), history of hemoptysis (more than 5ml fresh bleeding within 4 weeks);
* Corneal diseases of clinical significance. There is a history of retinal pigment epithelial detachment or evidence of the presence of retinal pigment epithelial detachment. History of age-related macular degeneration or evidence of age-related macular degeneration exists；
* Subjects with impaired cardiac function or heart disease of clinical significance;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limited toxicity (DLT) | 1 year
  To identify the dose-limited toxicity (DLT).
Maximum tolerated dose (MTD) | 1 year
  To identify the maximum tolerated dose (MTD).
Recommended Phase II Dose (RP2D) | 1 year
  To identify the Recommended Phase II Dose (RP2D).

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 2 year
  To preliminarily evaluate the AUC in patients with advanced solid tumors.
Peak Plasma Concentration (Cmax) | 2 year
  To preliminarily evaluate Cmax in patients with advanced solid tumors.
Time of peak plasma concentration (Tmax) | 2 year
  To preliminarily evaluate Tmax in patients with advanced solid tumors.
Overall response rate (ORR) | 2 year
  To preliminarily evaluate ORR in patients with advanced solid tumors.
Duration of Response (DoR) | 2 year
  To preliminarily evaluate DoR in patients with advanced solid tumors.
Median progression free survival (PFS) | 2 year
  To preliminarily evaluate PFS in patients with advanced solid tumors.
Median overall survival (OS) | 2 year
  To preliminarily evaluate OS in patients with advanced solid tumors.
Gene status | 2 year
  FGFR1-4, VEGFA, CSF1, CSF1R and other related gene status

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- CSPC ZhongQi Pharmaceutical Technology Co., Ltd., Beijing, China